CLINICAL TRIAL: NCT04127994
Title: Effect on Glycemic Variability, Weight and Oxidative Stress Markers FGF 21 in a Low Calorie Diet of Three Meals Compared With a Conventional Low Calorie Plan of Six Meals in Patients With Type 2 Diabetes With Overweight or Obesity
Brief Title: Glycemic Variability Comparing Two vs Six Meals in Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Miguel Ángel Gómez Sámano, MD, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2100
Record Dates: First submitted 2019-09-11; First posted 2019-10-16 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus Type 2; Overweight and Obesity; Meal Time
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 meals (Experimental): Patients with type 2 diabetes will be submitted to a 3 meal regimen for 3 months.
  We will compare their basal complete blood chemistry, somatometric measurements versus the same variables after 3 months.
  Interventions: Other: Comparing 3 versus 6 meals in type 2 diabetes patients
- 6 meals (Experimental): Patients with type 2 diabetes will be submitted to a 6 meal regimen for 3 months.
  We will compare their basal complete blood chemistry, somatometric measurements versus the same variables after 3 months.
  Interventions: Other: Comparing 3 versus 6 meals in type 2 diabetes patients

INTERVENTIONS:
Other: Comparing 3 versus 6 meals in type 2 diabetes patients — We will compare a 3 meals regimen versus a 6 meal regimen in patients with type 2 diabetes and overweight or obesity, to analyze which of the regimens have better outcomes in glycemic variability

SUMMARY:
The frequency of meals is a very important aspect of nutrition, with profound effects on human health and in life expectancy. Excessive energy consumption is totally associated with a significant increase in the incidence of chronic diseases including diabetes. That is why nutritional therapy is recommended for all people with diabetes mellitus type 1 and 2 as an effective complement to your medical treatment. For overweight or obese type 2 diabetic patients, a low-calorie diet along with healthy eating patterns are recommended for weight loss. Similarly, modest body weight decrease may provide clinical benefits in patients, such as improved blood glucose, blood pressure, lipid profile, and others. Data about the role of nutritional habits and energy density being important precursors of obesity and diabetes are well known. On the other hand, data regarding frequency and timing of meals and how these factors relate to corporal weight are not totally understood.

DETAILED DESCRIPTION:
In general, hypocaloric plans for patients with type 2 diabetes mellitus are consumed in five or six small meals per day. Eating more often is presumed to reduce hunger and thus energy consumption. However, the effects of meal frequency on human health and longevity are unclear.

Therefore, this study will be carried out in which the differences in the impact of nutritional therapy between a hypocaloric conventional 6 times meal versus a 3-meal low-calorie plan will be demonstrated.

The procedures will be as follows:

50 patients with DM2 from the Institute's Diabetes Clinic who are overweight or obese and between 40 and 70 years of age and who are found to have oral hypoglycemic agents, HbA1c less than 9% and less than 10 years old will be recruited of evolution.

Clinical evaluation:

A complete medical history and physical examination will be performed in order to confirm the presence of the inclusion criteria and rule out the presence of exclusion criteria. An anthropometric and body composition assessment (waist and hip circumference, height, weight and percentage of fat) as well as blood pressure measurement will be made. A history of coronary heart disease, menopausal status and use of hormone therapy, smoking, alcohol consumption and physical activity (through a questionnaire of physical activity validated in the Mexican population) will be conducted.

Nutritional assessment:

Patients will be divided into 2 groups without any distinction.

The first group of 25 patients will undergo a caloric restriction with a caloric restriction of 15% of their usual daily intake with a 40% macronutrient distribution in Carbohydrates, 20% Protein and 40% Lipids in three times of (TC6) over a period of 12 weeks in which the following variables will be measured: (Weight, Glucose Variability: Monitor, HbA1c, blood glucose, Lipid Profile, Oxidative stress, FGF-21, Blood Pressure and Hunger-Satiety Levels.)

At the first visit, the clinical evaluation will be elaborated, which consists of a complete physical examination in which vital signs will be measured, neck and head examination, examination of the thorax and abdomen, exploration of upper and lower extremities. As well as a complete nutritional assessment that includes; Assessment of body composition using bioimpedance with body composition analyzer jawon iOi 353, Reminder of food consumption of 72hrs to collect information on the diet of each patient. Based on the information collected will proceed to prescribe the individualized TC6 plan and will be given a 24/7 reminder format to be filled by the patient for a week, in addition to giving the indication to perform home glucose measurement once a day In random scheme.

To evaluate attachment to the nutritional plan, the patient will be cited 15 days later to perform daily consumption assessment using the 24/7 reminder format filled out by the patient and a 72hrs reminder performed through an interview. Likewise, levels of Hunger-Satiety will be measured with the tables of the institute Joslin validated for Mexican population.

If the patient adheres to the diet, blood samples will be taken for the measurement of the variables (HbA1C, Glucose, Lipid Profile, Insulin, FGF-21) and after that place the Medtronic model Ipro2 continuous glucose monitor with In order to monitor the patient's blood glucose for 7 days.

At the end of the 7 days, the patient will be asked to remove the sensor and re-evaluate dietary attachment.

The TC6 plan will be continued for 6 weeks, and at the end of this period the patient will be recalled to re-perform blood samples to measure the variables (HbA1C, Glucose, Lipid Profile, Insulin, FGF-21) Blood pressure and levels of Hunger-Satiety.

The TC6 regimen will be continued for a further 6 weeks. At the end of the period the patient will be asked to re-perform blood samples to measure the variables (HbA1C, Glucose, Lipid Profile, Insulin, FGF-21), Weight, Blood Pressure and Hunger-Satiety levels.

The second group of 25 patients will undergo a caloric restriction with a caloric restriction of 15% of their usual daily intake, with a 40% macronutrient distribution in Carbohydrates, 20% Protein and 40% Lipids in three times of (TC3) over a period of 12 weeks in which the following variables (Weight, Glucose Variability: Monitor, HbA1c, blood glucose, Lipid Profile, Oxidative, FGF-21, Blood Pressure and Hunger-Satiety levels are measured.) At the first visit, the clinical evaluation will be elaborated, which consists of a complete physical examination in which vital signs will be measured, neck and head examination, examination of the thorax and abdomen, exploration of upper and lower extremities. As well as a complete nutritional evaluation that includes, assessment of body composition using bioimpedance with jawon iOi 353 body composition analyzer, food consumption reminder of 72hrs to collect information on each patient's diet. Based on the information collected will proceed to prescribe the individualized TC3 plan and will be given a 24/7 reminder format to be filled by the patient for a week, in addition to giving the indication to perform home glucose measurement once a day in random scheme.

To evaluate attachment to the nutritional plan, the patient will be cited 15 days later to perform daily consumption assessment using the 24/7 reminder format filled out by the patient and a 72hrs reminder performed through an interview. Likewise, levels of Hunger-Satiety will be measured with the tables of the institute Joslin validated for Mexican population.

If the patient adheres to the diet, blood samples will be taken for the measurement of the variables (HbA1C, Glucose, Lipid Profile, Insulin, FGF-21) and after that place the Medtronic model Ipro2 continuous glucose monitor with in order to monitor the patient's blood glucose for 7 days.

At the end of the 7 days, the patient will be asked to remove the sensor and re-evaluate dietary attachment.

The TC3 plan will be continued for 6 weeks, and at the end of this period the patient will be recalled to re-perform blood samples to measure the variables (HbA1C, Glucose, Lipid Profile, Insulin, FGF-21) Blood pressure and levels of Hunger-Satiety. The TC3 regimen will be continued for a further 6 weeks. At the end of the period the patient will be asked to re-perform blood samples to measure the variables (HbA1C, Glucose, Lipid Profile, Insulin, FGF-21), Weight, Blood Pressure and Hunger-Satiety levels.

ELIGIBILITY:
Inclusion Criteria:

* Oral hypoglycemic agents
* HbA1c <9%
* Less than 10 years of evolution
* Diabetes Mellitus type 2
* Overweight or obese
* Age 40-70 years
* BMI ≥25 to < 40 kg/m

Exclusion Criteria:

* Obesity 3rd grade
* DM 1
* Hospitalization in the last 3 months
* >10 years of evolution
* HbA1c >9%
* Pregnancy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-08-17 (Actual); Primary Completion 2023-10-11 (Estimated); Study Completion 2023-10-11 (Estimated)

PRIMARY OUTCOMES:
Impact of 3 stroke diet in glycemic variability compared to a 6 stroke diet | 12 weeks
  Patients from both groups (3 stroke and 6 stroke diet) will be monitored for 7 days using intensive capillar blood glucose measurements 4 times per day (Fasting, 2 hours post breakfast, 2 hours post meal and 2 hours post dinner). The basal intensive blood glucose meaasurement monitoring will start at week 1 (first visit), and will end at day 7 and final intensive blood glucose meaasurement monitoring will start at week 11 and will end 7 days after (final visit) comparing glycemic variability between them. Mean difference of glycaemic variability (MAGE) calculated in mmol/L.

SECONDARY OUTCOMES:
Impact of 3 stroke diet in glycosylated hemoglobin levels compared to a 6 stroke diet | 12 weeks
  Mean difference of glycosylated hemoglobin represented in %
Impact of 3 stroke diet in fasting glucose levels compared to a 6 stroke diet | 12 weeks
  Mean difference of fasting glucose represented in mg/dL
Impact of 3 stroke diet in triglycerides levels compared to a 6 stroke diet | 12 weeks
  Mean difference of triglycerides represented in mg/dL
Impact of 3 stroke diet in cholesterol levels compared to a 6 stroke diet | 12 weeks
  Mean difference of cholesterol levels represented in mg/dL
Impact of 3 stroke diet in fibroblast growth factor 21 levels compared to a 6 stroke diet | 12 weeks
  Mean difference of fibroblast growth factor 21 levels represented in pg/ml.
Impact of 3 stroke diet in systolic and diastolic blood pressure compared to a 6 stroke diet | 12 weeks
  Mean difference of systolic and diastolic blood pressure represented in mmHg
Impact of 3 stroke diet in satiety compared to a 6 stroke diet | 12 weeks
  Mean difference of satiety will be estimated using hunger-satiety questionnaire (1-10 points)
Impact of 3 stroke diet in weight loss compared to a 6 stroke diet | 12 weeks
  Mean difference of weight represented in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel Gómez Sámano, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán ''INCMNSZ'', Mexico City, Mexico

DOCUMENTS (2):
  • Study Protocol (2017-01-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT04127994/Prot_001.pdf
  • Informed Consent Form (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT04127994/ICF_000.pdf